CLINICAL TRIAL: NCT00138970
Title: Randomised, Double-Arm, Controlled, Open-Label Study Comparing Calcineurin Inhibitor-Free Immunosuppression (Zenapax®, CellCept® and Prednisolone) and Cyclosporine A Based Immunosuppression (Sandimmun Neoral®, CellCept® and Prednisolone) on the Outcome of Renal Function and Acute Rejection in 0 DR Mis-Matched Renal Allograft Recipients
Brief Title: Calcineurin Inhibitor-Free Immunosuppression in Renal Transplant Recipients at Low Immunogenic Risk
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Oslo School of Pharmacy (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CLARIFI
Record Dates: First submitted 2005-08-29; First posted 2005-08-30 (Estimated); Last update posted 2005-12-01 (Estimated); Status verified 2005-08

CONDITIONS: Renal Transplant Recipients
Keywords: Cadaveric donor; Calcineurine free
MeSH Terms: interventions — Daclizumab; Mycophenolic Acid; Prednisolone; Cyclosporine

INTERVENTIONS:
Drug: Zenapax®, CellCept® and prednisolone
Drug: Sandimmun Neoral®, CellCept® and prednisolone

SUMMARY:
To compare renal function (51Cr-EDTA clearance) 12 months posttransplant, in primary renal allograft recipients (from cadaveric donor) at low immunogenic risk, 0 DR mis-match, receiving immunosuppressive therapy with A) Zenapax® (5 doses), CellCept® (1.5 g bid., aiming for TDM for total trough concentrations of 2-6 mg/L) and prednisolone or B) Sandimmun Neoral® (full dose), CellCept® (1.0 g bid.) and prednisolone.

DETAILED DESCRIPTION:
Primary Objective To compare renal function (51Cr-EDTA clearance) 12 months posttransplant, in primary renal allograft recipients (from cadaveric donor) at low immunogenic risk, 0 DR mis-match, receiving immunosuppressive therapy with A) Zenapax® (5 doses), CellCept® (1.5 g bid., aiming for TDM for total trough concentrations of 2-6 mg/L) and prednisolone or B) Sandimmun Neoral® (full dose), CellCept® (1.0 g bid.) and prednisolone.

Secondary Objectives To compare the two treatment groups with regard to: patient and graft survival (12 months), biopsy-proven and presumptive rejection episodes (3 and 12 months), posttransplant (12 months) incidence and severity of hypertension, hyperlipidemia, glucose intolerance, incidence of infection and tolerability and "success rate" of TDM guided CellCept® dosing in a calcineurin inhibitor-free immunosuppressive protocol over 12 months.

ELIGIBILITY:
Inclusion Criteria:

* 1. Patients of either gender above 18 years of age. 2. Patients who are recipients of primary, 0 DR mis-matched renal allografts from cadaveric donors (aged between 10 and 70 years).

  3. Patients who are single organ recipients (kidney only). 4. If the patients are women of childbearing potential, they must use safe contraceptives.

  5. Patients not previously treated with Zenapax® or Simulect®. 6. Patients must be capable to understand the information given about the study, including purpose and risks, and they must sign a statement of informed consent in accordance with the Helsinki declaration.

  7. Patients with white blood count greater than 2.5 x 109 /L (IU), platelet count greater than 100 x 109 /L (IU) or haemoglobin greater than 6 g/dL at the time of entry into the study.

Exclusion Criteria:

* 1. Patients who are recipients of HLA-identical renal transplants. 2. PRA positive (>20%) patients at any time the alst 6 months. 3. Patients who are unable to stay outside hospital as outpatients for 3 months.

  4. Patients who are unable to receive oral medication. 5. Patients with active peptic ulcer disease. 6. Patients with active infection. 7. Patients with disorders which might interfere with their ability to absorb oral medication, such as severe diarrhoea or patients with previously diagnosed diabetic gastroenteropathy.

  8. Patients who are pregnant or nursing mothers. 9. Patients with ongoing malignancies, excluding adequately treated skin carcinoma.

  10. Patients not able to adhere to the investigational immunosuppressive therapy.

  11. Patients receiving bile-acid sequestants.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70
Dates: Start 2002-01; Study Completion 2005-02

PRIMARY OUTCOMES:
The primary efficacy endpoint is the renal function, evaluated by 51Cr-EDTA clearance and normalized for 1.73 m2 body-surface, at 12 months posttransplant.

SECONDARY OUTCOMES:
• Combined patient and graft survival at 12 months posttransplant.
• Proportion of patients with biopsy-proven acute rejection or acute rejection (biopsy proven + presumptive) episode at 3 and 12 month posttransplant.
• Incidence and severity of hypertension at 10 weeks and 12 months posttransplant.
• Incidence and severity of dyslipidemia at 10 weeks and 12 months posttransplant.
• Incidence of glucose intolerance at 10 weeks and 12 months posttransplant.
• Incidence of treatment failure at 12 months posttransplant.
• Success rate of TDM guided CellCept® dosing at 3 months posttransplant.
• Infection rate.

CONTACTS AND LOCATIONS:
Overall Officials: Anders Hartmann, MD, Principal Investigator — Rikshospitalet, Section of Nephrology